CLINICAL TRIAL: NCT05406830
Title: Evaluating the Efficacy of Acupuncture for Patients With Asymptomatic Hyperuricemia (HUA): A Multicenter Randomized Controlled Clinical Trial
Brief Title: Efficacy Study of Acupuncture on Asymptomatic Hyperuricemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lingling Yu (103250) (Other)
Collaborators: Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other); Xianning Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Lingling Yu (103250), Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021HUATJ01
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Asymptomatic Hyperuricemia
Keywords: Manual Acupuncture; Asymptomatic Hyperuricemia; Serum Uric Acid; Efficacy; Safety

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum acupuncture (VA) (Experimental): Participants will be treated by real manual acupuncture and usual care. They will be treated twice a week for 8 weeks, to fulfill a 16-session treatment course. Each acupuncture treatment session for patients will be 30 minutes in duration.
  Interventions: Device: verum acupuncture; Behavioral: health education
- Sham acupuncture (SA) (Sham Comparator): Participants will be treated by non-penetrating sham acupuncture and usual care. They will be treated twice a week for 8 weeks, to fulfill a 16-session treatment course. Each acupuncture treatment session for patients will be 30 minutes in duration.
  Interventions: Behavioral: health education; Device: sham acupuncture

INTERVENTIONS:
Device: verum acupuncture — The special type of acupuncture needles will be inserted into the skin of standard acupuncture points and manipulated manually by using the techniques such as lifting, thrusting, and twirling, until the internal compound sensation known as deqi.
  Arms: Verum acupuncture (VA)
Behavioral: health education — According to the Multidisciplinary Expert Consensus on the Diagnosis and Treatment of Hyperuricemia related Diseases in China and the 2012 Guidelines of the American College of Rheumatology, health education should be given as basic prevention. These include weight control, regular exercise, limiting alcohol and high-purine and high-fructose diets, encouraging dairy and fresh vegetables and drinking moderate amounts of water, and not recommending or limiting soy products.
Device: sham acupuncture — We will use a non-insertive sham control. Sham points are located at 5 cun lateral to the seventh, eighth, ninth, tenth, eleven and twelve thoracic spine. Cun is a distance measure unit used in locating acupoints in traditional Chinese medicine (TCM) acupuncture, and the width of patient's thumb interphalangeal joint is regarded as one cun.
  Arms: Sham acupuncture (SA)

SUMMARY:
hyperuricemia (HUA) is an important risk factor for various chronic diseases, such as gout, and the current treatment programs for HUA are not ideal. It is urgent to find new methods to prevent and treat HUA and to carry out early clinical intervention. Acupuncture is commonly used for the treatment of HUA, while the evidence for its efficacy is still uncertain. This clinical trial aimed to evaluate the efficacy and safety of manual acupuncture for asymptomatic HUA.

DETAILED DESCRIPTION:
This is a multicentre, stratified, randomized, sham-controlled clinical trial. 180 eligible participants will be randomly allocated into verum acupuncture group or sham acupuncture group, in a 1:1 ratio. The verum acupuncture group will receive 16 sessions of manual acupuncture treatments over an eight-week period, while the sham acupuncture group will receive sham acupuncture treatments with non-penetrating needling. Health education will be provided to participants in the two groups. The primary outcomes will be the changes in the mean levels of serum uric acid 8 weeks after randomization. The secondary outcomes will be the changes in the mean levels of serum uric acid 4, 12, 16, and 20 weeks after randomization. Other secondary outcomes included effective rates, the proportion of patients with acute gouty arthritis, changes in body weight and BMI, safety evaluation and deqi evaluation. The central randomization and data collection will be conducted by an electronic data management system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as hyperuricemia; and
* Fasting blood uric acid level ≥ 7-11.0 mg/dL after 1 month of low-purine diet; and
* Without history of gouty arthritis; and
* Without drug treatment for hyperuricemia or stop uric acid-lowering drug treatment ≥12 weeks; and
* 18.5kg/m2≤BMI≤30.0kg/ m2; and
* Able to signing a informed consent.

Exclusion Criteria:

* Those who are using or have used one of the following drugs for the treatment of hyperuricemia 12 weeks before eligibility evaluation, such as: allopurinol, benzbromarone, probesulfan, bugelone, toppirosteine, Busotan; and
* Patients are using or used other drugs that affect uric acid metabolism in the past 12 weeks, such as: thiazide diuretics, angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, compound reserpine, pyrazinamide, nitrates fendipine, propranolol, and benzbromarone; and
* Patients have history of gouty arthritis; and
* Combined with secondary hyperurmicema, such as bone marrow and lymphoproliferative diseases, tumor radiotherapy and chemotherapy, liver cirrhosis and drug-induced hyperurmicema; and
* Combined with one of the following comorbidities: hypertension, diabetes, stroke, coronary heart disease, severe liver and kidney damage (≥CKD stage 2, or high creatinine, urea, glutamate, glutamate ≥ 2 times of the limit of clinical normal values); and
* Combined with severe neuropsychological diseases, such as severe anxiety, depression, and intellectual disability; and
* Pregnant women; and
* Unwilling to accept acupuncture treatment; and
* Illiterate, or patients unable to sign informed consent; and
* The completion rate of baseline screening data is ≤80%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the mean level of serum uric acid from baseline. | At baseline, and at 8 weeks after randomization.
  The changes in the mean level of serum uric acid at 8 weeks after randomization compared to baseline

SECONDARY OUTCOMES:
Changes in the mean level of serum uric acid from baseline. | At baseline, at 4, 12, 16, and 20 weeks after randomization.
  The changes in the mean level of serum uric acid at 4, 12, 16, 20 weeks after randomization compared to baseline
Effective rate of patients with serum uric acid ≤ 6.0 mg/dL | 4, 8, 12, 16 and 20 weeks after randomization
  The ratio of patients with serum uric acid ≤ 6.0 mg/dL at weeks 4, 8, 12, 16 and 20 after randomization
Effective rate of patients with serum uric acid ≤ 7.0 mg/dL | 4, 8, 12, 16 and 20 weeks after randomization
  The ratio of patients with serum uric acid ≤ 7.0 mg/dL at weeks 4, 8, 12, 16 and 20 after randomization
The proportion of patients with acute gouty arthritis | Weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The proportion of patients with acute gouty arthritis per 4-week cycle after randomization.
Changes in body weight of patients | 4, 8, 12, 16 and 20 weeks after randomization
  Changes in body weight of patients at 4, 8, 12, 16, and 20 weeks after randomization.
Changes in the dose of intake of acute medication. | Weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the dose of intake of acute medication per 4-week cycle after randomization.
Arrival of qi assessment | Immediately following each session of acupuncture treatment.
  The Chinese Version of the Massachusetts General Hospital Acupuncture Sensation Scale Acupuncture sensations will be measured by the Massachusetts General Hospital (MGH) Acupuncture Sensation Scale (MASS)
Safety evaluation | Immediately following each session of acupuncture treatment.
  Adverse events during the acupuncture process

OTHER OUTCOMES:
60-item NEO Personality Inventory-Short Form (NEO-FFI) | At baseline only once.
Chinese medicine constitution classification | At baseline only once.
Acupuncture Expectancy Scale | At baseline only once.
Change in Beck Anxiety Inventory(BAI). | At baseline only once.
Change in Beck Depression Inventory II(BDI- II). | At baseline only once.
Change in Patient-Doctor Relationship Questionnaire(PDRQ-9) . | At baseline only once.
Change in Difficult Doctor-Patient Relationship Questionnaire(DDPRQ-10). | At baseline only once.

CONTACTS AND LOCATIONS:
Overall Officials: Shenghao Tu, PhD, Principal Investigator — Institute of Integrated Traditional Chinese and Western Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan,430030, China
Locations (1):
- Institute of Integrated Traditional Chinese and Western Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Yu LL, Li CN, Fang MY, Ma Y, Wang B, Lin FP, Liu WH, Tu SH, Chen Z, Xie WX, Zhang RY, Huang Y, Zheng CH, Wang Y. Evaluating the effectiveness and safety of acupuncture on serum uric acid in asymptomatic hyperuricemia population: a randomized controlled clinical trial study protocol. Front Endocrinol (Lausanne). 2023 Oct 13;14:1218546. doi: 10.3389/fendo.2023.1218546. eCollection 2023. PMID 37900149